CLINICAL TRIAL: NCT00682227
Title: Phase I Study of Peptide Vaccination Therapy Using Novel Cancer Testis Antigens for Locally Advanced, Recurrent, or Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: Peptide Vaccination in Treating Patients With Esophageal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Yamanashi (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Koji Kono, First Department of Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMU-01
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Esophageal Cancer
Keywords: Epitope peptide, CTL, Esophageal cancer, Vaccination
MeSH Terms: conditions — Esophageal Neoplasms | interventions — LY6K protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: TTK, LY6K, and IMP-3 peptides

INTERVENTIONS:
Biological: TTK, LY6K, and IMP-3 peptides — Each of three peptides (1mg) mixed with IFA (1ml) were injected every week at five round.

SUMMARY:
The purpose of this study is to evaluate the safety and immunological monitoring for peptide vaccination therapy using novel cancer testis antigens for locally advanced, recurrent, or metastatic esophageal squamous cell carcinoma

DETAILED DESCRIPTION:
We recently identified three HLA-A2402-restricted epitope peptides (TTK protein kinase (TTK), lymphocyte antigen 6 complex locus K (LY6K), and insulin-like growth factor (IGF)-II mRNA binding protein 3 (IMP-3)) derived from novel Cancer-Testis antigens (CTA) for the development of immunotherapies against esophageal squamous cell carcinoma (ESCC), and reported that the pre-existence of specific T cell responses to these epitope peptides were frequently seen in ESCC patients. Then, we performed Phase I vaccination trial using multi-epitopes involving TTK, LY6K, and IMP-3 peptides for locally advanced, recurrent or metastatic esophageal squamous cell carcinoma who had failed for the standard therapy. Each of three HLA-A2402-restricted epitope peptides mixed with IFA were injected every week at five round. Primary endpoints were to evaluate the safety and feasibility of the therapy. Secondary endpoints were to investigate the immunological monitoring and clinical effect.

ELIGIBILITY:
Inclusion Criteria:

* DISEASE CHARACTERISTICS 1. Locally advanced, recurrent or metastatic esophageal squamous cell carcinoma who had failed for the standard therapy

PATIENTS CHARACTERISTICS

1. ECOG performance status 0-2
2. Age≧20 years, 80≦years
3. WBC≥ 2,000/mm³ Platelet count ≥ 75,000/mm³ Total bilirubin ≤ 2.0 x the institutional normal upper limits AST, ALT, ALP ≤ 2.5 x the institutional normal upper limits Creatinine ≤ 1.5 x the institutional normal upper limits
4. Patients must be HLA-A2402
5. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Pregnancy (women of childbearing potential: Refusal or inability to use effective means of contraception)
2. Breastfeeding
3. Serious bleeding disorder
4. Serious infections requiring antibiotics
5. Concomitant treatment with steroids or immunosuppressing agent
6. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Safety (toxicities as assessed by NCI CTCAE version 3) | 3 months

SECONDARY OUTCOMES:
Immunological and clinical response | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Koji Kono, MD.PhD, Principal Investigator — First Depatment of Surgery
Locations (1):
- University of Yamanashi, First Department of Surgery, 1110 Shimokato, Chuo-city, Yamanashi, Japan

REFERENCES:
- [Background] Lin YM, Furukawa Y, Tsunoda T, Yue CT, Yang KC, Nakamura Y. Molecular diagnosis of colorectal tumors by expression profiles of 50 genes expressed differentially in adenomas and carcinomas. Oncogene. 2002 Jun 13;21(26):4120-8. doi: 10.1038/sj.onc.1205518. PMID 12037668
- [Background] Hasegawa S, Furukawa Y, Li M, Satoh S, Kato T, Watanabe T, Katagiri T, Tsunoda T, Yamaoka Y, Nakamura Y. Genome-wide analysis of gene expression in intestinal-type gastric cancers using a complementary DNA microarray representing 23,040 genes. Cancer Res. 2002 Dec 1;62(23):7012-7. PMID 12460921
- [Background] Suda T, Tsunoda T, Daigo Y, Nakamura Y, Tahara H. Identification of human leukocyte antigen-A24-restricted epitope peptides derived from gene products upregulated in lung and esophageal cancers as novel targets for immunotherapy. Cancer Sci. 2007 Nov;98(11):1803-8. doi: 10.1111/j.1349-7006.2007.00603.x. PMID 17784873
- [Background] Ishikawa N, Takano A, Yasui W, Inai K, Nishimura H, Ito H, Miyagi Y, Nakayama H, Fujita M, Hosokawa M, Tsuchiya E, Kohno N, Nakamura Y, Daigo Y. Cancer-testis antigen lymphocyte antigen 6 complex locus K is a serologic biomarker and a therapeutic target for lung and esophageal carcinomas. Cancer Res. 2007 Dec 15;67(24):11601-11. doi: 10.1158/0008-5472.CAN-07-3243. PMID 18089789
- [Derived] Kono K, Mizukami Y, Daigo Y, Takano A, Masuda K, Yoshida K, Tsunoda T, Kawaguchi Y, Nakamura Y, Fujii H. Vaccination with multiple peptides derived from novel cancer-testis antigens can induce specific T-cell responses and clinical responses in advanced esophageal cancer. Cancer Sci. 2009 Aug;100(8):1502-9. doi: 10.1111/j.1349-7006.2009.01200.x. Epub 2009 May 14. PMID 19459850